CLINICAL TRIAL: NCT00437996
Title: Epidural Analgesia During Labour. Impact of Clonidine Addition to Levobupivacaine and Sufentanil
Brief Title: Comparative Affect of a Continuous Epidural Infusion of Clonidine During Labour. Prospective Double Blind Randomized Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2006.424
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Normal Pregnancy
Keywords: Labor analgesia - clonidine - epidural
MeSH Terms: interventions — Clonidine; Levobupivacaine; Sufentanil

INTERVENTIONS:
Drug: Clonidine
Drug: Levobupivacaine
Drug: Sufentanil

SUMMARY:
Addition of clonidine to an epidural mixture of local anaesthetic and morphine improves analgesia and reduces the frequency of motor blockade during epidural analgesia. several side effects are possible mostly somnolence and hypotension. Association of continuous clonidine infusion with low concentrations of levobupivacaïne and sufentanil was not studied during labour. The objective of this study is to compare the effectiveness and the side effects of a PCEA with levobupivacaïne 0,0625 % and sufentanil 0.25 microg.ml-1, without addition of clonidine, and with addition of clonidine at a concentrations of 2 microg.ml-1.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA class I or II
* Variable parity
* Aged of 18 years or more
* With a normal pregnancy
* Cervical dilation between 3 and 8 cm)
* Wishing an epidural analgesia
* Normal childbirth
* Giving their written assent
* Affiliated with a social security system
* Must have had an anaesthesia consultation more than 48 hours before inclusion.

Exclusion Criteria:

* Request of the patient
* Failure of epidural analgesia
* Childbirth in the 90 minutes following the induction of analgesia
* Realization of a Caesarean section

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-02; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Score of quality at the time of the childbirth based on a 4-point scale : motor blockade - no sensation - nonpainful sensation - pain.

SECONDARY OUTCOMES:
Motor blockade quantification by a score of modified Bromage specific way.
Labor analgesia.
Circulatory parameters(arterial pressure and heart rate will be noticed at 5 - 10 - 15 - 20 - 30 - 60 minutes and every hour until childbirth).

CONTACTS AND LOCATIONS:
Overall Officials: HENRI-JACQUES CLEMENT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Henri Jacques CLEMENT, Lyon
  - Anesthesie Reanimation - Gynecologie - Hopital de La Croix Rousse, Lyon

REFERENCES:
- [Derived] Wallet F, Clement HJ, Bouret C, Lopez F, Broisin F, Pignal C, Schoeffler M, Derre E, Charpiat B, Huissoud C, Aubrun F, Viale JP. Effects of a continuous low-dose clonidine epidural regimen on pain, satisfaction and adverse events during labour: a randomized, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2010 May;27(5):441-7. doi: 10.1097/EJA.0b013e3283365944. PMID 20299988